CLINICAL TRIAL: NCT05630209
Title: A Safety and Feasibility Study to Evaluate Blood Brain Barrier Disruption Using Exablate MR Guided Focused Ultrasound in Combination With Doxorubicin in Treating Pediatric Patients With Diffuse Intrinsic Pontine Gliomas (DIPG)
Brief Title: Blood Brain Barrier (BBB) Disruption Using Exablate Focused Ultrasound With Doxorubicin for Treatment of Pediatric Diffuse Intrinsic Pontine Gliomas (DIPG)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BT016
Record Dates: First submitted 2022-11-18; First posted 2022-11-29 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Brain Tumor
Keywords: DIPG; Focused Ultrasound; Chemotherapy; Phase I trial; Pediatrics
MeSH Terms: conditions — Brain Neoplasms | interventions — Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Blood Brain Barrier Disruption (BBBD) (Experimental): Exablate MR Guided Focused Ultrasound for Blood Brain Barrier Disruption with Doxorubicin for treating pediatric patients with DIPG
  Interventions: Device: Exablate; Drug: Doxorubicin

INTERVENTIONS:
Device: Exablate — Blood Brain Barrier Disruption (BBBD) via Exablate Type 2 system with microbubble resonators on the day of Doxorubicin infusion to treat DIPG brain tumors
  Other Names: Exablate BBBD
Drug: Doxorubicin — Doxorubicin infusion
  Other Names: Adriamycin; Rubex

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of targeted blood brain barrier disruption with Exablate Model 4000 Type2.0/2.1 in combination with Doxorubicin therapy for the treatment of DIPG in pediatric patients

DETAILED DESCRIPTION:
This is a prospective, single arm, non-randomized feasibility study to evaluate the safety, feasibility and preliminary efficacy of Blood Brain Barrier Disruption (BBBD) using the Exablate Type 2 system in pediatric patients with Diffuse Intrinsic Pontine Gliomas (DIPG) undergoing Doxorubicin chemotherapy. The study will be conducted at up to three sites in the United States. Patients will undergo 3 treatment cycles, approximately 4-6 weeks apart. The study aims to establish feasibility and safety of Exablate BBBD in conjunction with Doxorubicin in the treatment of pediatric DIPG and assess preliminary efficacy in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 21 years, inclusive. Subjects younger than 5 years old may be eligible after discussion with the Sponsor Medical Monitor/designee (i.e. DSMB).
* Patient diagnosed with DIPG
* At least 4-week and not greater than 12 weeks from completion of radiation therapy
* Post-radiation imaging does not show evidence of necrosis/ hemorrhage or other features that contraindicate MRgFUS
* If brain surgery occurred, at least 14 days passed since last brain surgery and the patient is fully recovered and neurologically stable
* If on steroids, stable or decreasing dose for at least 7 days prior to study entry
* Stable or improving neurologic status for 7 days prior to study entry
* Able and willing to give consent and/or assent or have a legal guardian who is able and willing to do so
* Able to attend all study visits and with life expectancy of at least 6 months

Exclusion Criteria:

* Tumor not visible on any pre-therapy or post-radiation imaging
* Previous participation in other chemotherapy, molecularly targeted therapy, or immunotherapy treatment-related phase 1 or 2 trials
* Symptoms and signs of increased intracranial pressure
* Subject with metastatic disease
* Subject with ventricular peritoneal shunt
* Subject receiving bevacizumab (Avastin) therapy or increasing doses of steroids
* Anti-coagulant therapy, or medications known to increase risk of hemorrhage, (e.g., ASA, non-steroidal anti-inflammatory drugs [NSAIDs], statins) within washout period prior to treatment
* History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage.
* Hypertension per age
* Cerebral or systemic vasculopathy, including intracranial thrombosis, vascular malformation, cerebral aneurysm, or vasculitis
* Immunosuppression (corticosteroids to prevent/treat brain edema are permitted).
* Patients with positive HIV status
* Active seizure disorder or epilepsy (seizures despite medical treatment) for a minimum of 4 weeks prior to first cycle/Exablate BBBD procedure captured by history
* Known sensitivity to gadolinium-based contrast agents
* Known sensitivity to DEFINITY® ultrasound contrast agent or known hypersensitivity to perflutren microsphere or its components, e.g., polyethylene glycol
* Contraindication to Doxorubicin
* Previous treatment with complete cumulative doses of Doxorubicin, daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones
* Severely impaired renal function with estimated glomerular filtration rate <2 standard deviations for age
* Patients that may require trastuzumab during the study
* Patients that may require inhibitors and inducers of CYP3A4, CYP2D6, and/or P-gp during the study

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | 2 years
  All adverse events from first treatment to end of study will be documented and reported according to the CTCAE terminology and severity scale

SECONDARY OUTCOMES:
Blood Brain Barrier Disruption (BBBD) | immediately post BBBD sonication
  BBBD will be assessed as a comparative ratio measured in pre and post-sonication contrast-enhanced MR images

OTHER OUTCOMES:
Progression Free Survival (PFS) | 2 years
  PFS will be assessed based on the Response Assessment in Pediatric Neuro-Oncology (RAPNO) scale.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Cook Children's Health Care System, Fort Worth, Texas